CLINICAL TRIAL: NCT00859716
Title: A Randomized, Double-Blind, Placebo Controlled Vaccination-Challenge Study of ACE393 to Determine Efficacy Against the Symptoms of Moderate to Severe Campylobacter Jejuni Infection in Normal Healthy Volunteers
Brief Title: ACE393-103 Vaccination Challenge Study
Acronym: ACE393-103VC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TD Vaccines A/S (Industry)
Collaborators: SNBL Clinical Pharmacology Center, Inc. (Industry); Johns Hopkins University (Other); University of Vermont (Other); SGS U.S. Testing Company Inc. (Industry); Fulcrum Pharma (Europe) Ltd (Unknown)
Responsible Party: Ingelise Saunders/CEO, ACE BioSciences A/S
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACE393-103; BB013742
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Campylobacter Infection
Keywords: Vaccination; Diarrhea; Traveler's Diarrhea; Campylobacter jejuni; C. jejuni; Campylobacter; Campy
MeSH Terms: conditions — Campylobacter Infections; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): vaccination with ACE393 followed by challenge with campylobacter jejuni
  Interventions: Biological: ACE393
- 2 (Placebo Comparator): Placebo vaccination followed by challenge with campylobacter jejuni
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: ACE393 — ACE393 250 micrograms as intra muscular injection at day 0 and day 21
  Other Names: Campylobacter jejuni
  Arms: 1
Biological: Placebo vaccine — Placebo 500 micrograms Alhydrogel as intra muscular injection at day 0 and day 21
  Other Names: Campylobacter jejuni
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether ACE393 vaccination can protect against Campylobacteriosis in a challenge model.

DETAILED DESCRIPTION:
This study is a randomized, double blind, parallel group, placebo controlled study, in which subjects, with no evidence of prior C.jejuni infections or immunity, will be vaccinated with ACE393, a protein sub-unit vaccine, or placebo, and then subsequently challenged with C.jejuni. The study will include vaccination of approximately 72 subjects, with the aim of challenging a total of 60 subjects. ACE393 or placebo will be administered twice by intramuscular injection on an outpatient basis, three weeks apart and then the subjects will be challenged three weeks later with C.jejuni. During the inpatient monitoring period, volunteers will be evaluated daily for safety, clinical signs and symptoms of disease and stool microbiology). Criteria for early institution of oral hydration, intravenous fluids, serum electrolyte monitoring, blood cultures, and/or antibiotics are predefined. All volunteers will receive antibiotic therapy 6 days after challenge (unless treated early). Discharge criteria are predefined. Post-discharge follow-up will further monitor safety, confirm C .jejuni eradication after antibiotic therapy, and assess immunologic response.

ELIGIBILITY:
Inclusion criteria (selected):

* Male or female between 18 and 50 years of age.
* General good health, without significant medical illness, abnormal physical examination findings or clinical laboratory abnormalities as determined by the principal investigator or the principal investigator in consultation with the medical monitor and sponsor.
* Negative serum pregnancy test at screening.

Exclusion Criteria (selected):

* Immunosuppressive illness or clinically significant IgA deficiency.
* Positive serology results for HIV, HBsAg, or HCV antibodies.
* Evidence of inflammatory arthritis on examination and/or HLA-B27 positive.
* Allergy or prior intolerance to selected antibiotics (specified in the protocol)
* Fewer than 3 stools per week or more than 3 stools per day as the usual frequency; or passing of loose or liquid stools other than on an occasional basis.
* History of diarrhea.
* Stool culture positive for Campylobacter, other bacterial enteropathogens and intestinal parasites.
* History of microbiologically confirmed Campylobacter infection.
* History of vaccination for or ingestion of Campylobacter.
* Immunologic evidence of Campylobacter exposure
* Serologic evidence of prior Campylobacter infection.
* Cell mediated immune response evidence of prior Campylobacter infection.
* Fever within 48 hours preceding challenge.
* Presence of any signs or symptoms indicative of active infection.
* Diarrhea occurring in the 7 days prior to challenge.
* Stool culture positive for Campylobacter, other bacterial enteric pathogens or intestinal parasites.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-03 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Moderate or Severe Diarrhea | 20 weeks

SECONDARY OUTCOMES:
Median Total (individual) stool number (grade 3-5 stools, diarrheal episodes only) | 20 Weeks
Median Total (individual) stool volume (grade 3-5 stools, diarrheal episodes only) | 20 weeks
Maximum stool number and volume in a 24 hr period (grade 3-5 stools, diarrheal episodes only) | 20 weeks
Incidence of severe diarrhea | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, MD, Principal Investigator — Shin Nippon Biomedical Laboratories
Locations (1):
- Shin Nippon Biomedical Laboratories, Baltimore, Maryland, United States

REFERENCES:
- See also: Sponsor — http://www.acebiosciences.com